CLINICAL TRIAL: NCT02091726
Title: Phase 4 Field Trial of the Unicirc Instrument With Tissue Adhesive
Acronym: Unicirc003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simunye Primary Health Care (Other)
Responsible Party: Principal Investigator, Peter Millard, PI, Simunye Primary Health Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Unicirc 003
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Male Circumcision
Keywords: Circumcision; HIV prevention; Surgical device; Cyanoacrylate; Tissue Adhesive; voluntary
MeSH Terms: interventions — Cyanoacrylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unicirc with tissue adhesive (Experimental): Circumcision with Unicirc instrument, followed by wound sealing with cyanoacrylate
  Interventions: Procedure: Unicirc instrument plus cyanoacrylate tissue adhesive

INTERVENTIONS:
Procedure: Unicirc instrument plus cyanoacrylate tissue adhesive — Volunteers will be circumcised using the Unicirc surgical instrument and the incision will be sealed using cyanoacrylate tissue adhesive
  Other Names: Unicirc; Cyanoacrylate

SUMMARY:
This is a field trial of the Unicirc instrument to excise the foreskin, plus use of cyanoacrylate tissue adhesive to seal the wound.

ELIGIBILITY:
Inclusion Criteria:

* Men at least 18 years of age

Exclusion Criteria:

* Poor general health
* Anatomical abnormalities that would complicate circumcision
* Bleeding disorder
* Ongoing infection
* Cannot attend followup visits

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Goldstuck, MD, Study Director — Department of Obstetrics and Gynaecology, Tygerberg Hospital, Cape Town, South Africa
Locations (1):
- Simunye Primary Healthcare, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Millard PS, Goldstuck ND. No-needle, single-visit adult male circumcision with Unicirc: a multi-centre field trial. PLoS One. 2015 Mar 30;10(3):e0121686. doi: 10.1371/journal.pone.0121686. eCollection 2015. PMID 25822727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three generalist physicians (GPs) performed the circumcisions in individual consultation rooms in their own primary health care clinic.
  The study took place between January 20 and July 4, 2014.
Period: Overall Study
Arm/Group | Unicirc With Tissue Adhesive
Started | 110
1 Week Followup | 110
4 Week Followup | 104
Completed | 104
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Volunteers
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 110
Region of Enrollment [Number; unit: participants]
  South Africa | 110

OUTCOME MEASURES:

1. Primary Outcome: Time for Procedure
Description: Intraoperative time, total
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: Min
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 110
Min | 9.0 [9.0 to 10.0]

2. Secondary Outcome: Completely Healed at 4 Weeks
Description: Definition: Completely epithelialized; no superficial ulcerations or granulation tissue present
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 104
participants | 94

3. Secondary Outcome: Wound Separation
Description: Wound separation caused by adhesive failure (minor --requires no treatment)
Time Frame: 4 weeks
Population: Wound dehiscence < 2 cm. None required treatment. There were no participants with wound dehiscence > 2 cm.
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 110
participants
  Separation > 2 cm longitudinally | 0
  Separation < 2 cm longitudinally | 5

4. Secondary Outcome: Cosmetic Result Excellent
Description: Excellent: scar line straight without any irregularity Irregular: Some irregularity to scar line Scalloped: wavy appearane to scar line
Time Frame: 4 weeks
Population: 104 men came for their 4-week followup but the doctor(s) failed to note the cosmetic result in 2 men.
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 102
participants | 101

5. Secondary Outcome: Participant Fully Satisfied and Would Recommend to Friends and Family
Description: Yes to both of the following questions: Are you fully satisfied with your circumcision result? Would you recommend circumcision to friends or family?
Time Frame: 4 weeks
Population: 104 men came for their 4-week followup, but 1 man did not complete the satisfaction questions.
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive
Number analyzed (Participants) | 103
participants | 103

ADVERSE EVENTS:
Time Frame: Time period: 4 weeks
Description: Active followup of volunteers at 1 and 4 weeks
Arm/Group | Unicirc With Tissue Adhesive
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 7/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unicirc With Tissue Adhesive (N=110)
Bleeding requiring suture (Surgical and medical procedures) | 5 (5)
Infection requiring antibiotics (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No